CLINICAL TRIAL: NCT02648334
Title: Randomized Comparison of Drug-Coated Balloons for the Treatment of Superficial Femoral and Popliteal Peripheral Artery Disease: Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: Randomized Comparison of DCB for the Treatment of Superficial Femoral and Popliteal Peripheral Artery Disease
Acronym: DCB-SFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Whan Lee, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Seung-Whan Lee, M.D., Ph.D., Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2015-08
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Angioplasty, Balloon; Catheterization, Peripheral; Popliteal Artery; Femoral Artery
Keywords: Drug-Coated Balloon; Superficial Femoral artery; popliteal peripheral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IN.PACT drug coated balloon (Active Comparator): IN.PACT drug coated balloon
  Interventions: Device: IN.PACT drug coated balloon
- Lutonix drug coated balloon (Experimental): Lutonix drug coated balloon
  Interventions: Device: Lutonix drug coated balloon

INTERVENTIONS:
Device: IN.PACT drug coated balloon
  Arms: IN.PACT drug coated balloon
Device: Lutonix drug coated balloon
  Arms: Lutonix drug coated balloon

SUMMARY:
This study evaluates the safety and effectiveness Percutaneous Transluminal Angioplasty(PTA) using Drug-Coated Balloons for the treatment of Superficial Femoral and popliteal peripheral Artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and above
* Subject with claudication or critical limb ischemia(Rutherford classification level 2~5)
* Subject with total occlusion or stenosis ≥70%(de novo, restenosis)
* Vessel diameter 4~6mm
* Success to guide wire pass
* Patients who don't have known hypersensitivity or allergy for dual-platelets
* Willing and able to provide informed written consent

Exclusion Criteria:

* Acute stage
* Acute thrombosis in target limb or target vessel
* Failure to guide wire pass
* Distal outflow
* Lesion with poor inflow
* Life expectancy ≤ 2 years
* Allergic to paclitaxel
* Pregnant or breast feeding woman or disagree with contraception or having children

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
the event rate of composite event | 1 year
  all cause death, revascularization due to amputation or clinical evidence

SECONDARY OUTCOMES:
all cause death | 2 years
cardiac death | 2 years
myocardial infarction | 2 years
stroke | 2 years
amputation of target limb | 2 years
target lesion revascularization | 2 years
The change of Rutherford classification | 2 years
The change of ABI(ankle-brachial index) score | 2 years
MACE | 2 years
  major adverse cardiac event(death, myocardial infarction, stroke)
thrombosis | 2 years

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Hallym University Sacred Heart Hospital, Anyang
  - Gyeongsang National University Changwon Hospital, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Myongji Hospital, Goyang-si
  - Seoul national university Bundang hospital, Gyeonggi-do
  - Jesushospital, Jeonju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Veterans Hospital, Pusan
  - Chungnam National University Sejong Hospital, Sejong
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Veterans Hospital Service Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
This is not publicly funded trial.